CLINICAL TRIAL: NCT04197856
Title: Direct Letters to Relatives at Risk of Hereditary Cancer- a Multi-centre Randomised Controlled Trial of Healthcare-assisted Versus Family-mediated Risk Disclosure at Swedish Cancer Genetics Clinics (DIRECT-study)
Brief Title: Direct Information to At-risk Relatives
Acronym: DIRECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Göteborg University (Other); Lund University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Rosen, Principal investigator, MD, PhD, Specialist in Clinical genetics, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: The Swedish DIRECT study; 2018-00964 (Other Grant/Funding Number: Swedish Research council for health, worklife and welfare); 2020-1107 (Other Grant/Funding Number: Swedish Cancer Society); 2022-02226 (Other Grant/Funding Number: Swedish research council); 86719 (Registry Identifier: RCC Cancerstudier i Sverige (in Swedish))
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Familial Breast Cancer; Familial Colorectal Cancer; Hereditary Breast and Ovarian Cancer Syndrome; Hereditary Breast Cancer; Lynch Syndrome
Keywords: hereditary cancer risk; prevention; family-mediated disclosure; healthcare-assisted disclosure; information disclosure; risk information; genetic risk
MeSH Terms: conditions — Breast Cancer, Familial; Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Intervention Model Description: Multi-centre, parallel assignment, balanced ratio, investigator-blinded, randomised, controlled superiority trail in Sweden.
Masking Description: Since the intervention in this trial is an offer of sending physical direct letters to at-risk relatives, neither the health care providers nor the study participant can be blinded to the allocation. However, the final data analysis will be performed by a statistician blinded to the study arm allocations and subgroups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control / Family-mediated disclosure (standard care) (Active Comparator): Genetic counseling according to current clinical practice
  Interventions: Other: Standard care encouraging family-mediated disclosure of hereditary cancer risk
- Intervention / Health-care assisted disclosure (Experimental): Genetic counseling according to current clinical practice with the addition of an offer from health care provider to mail letters directly to eligible at-risk relatives.
  Interventions: Other: Standard care encouraging family-mediated disclosure of hereditary cancer risk; Other: Offer of health-care assisted disclosure by sending direct letters to at-risk relatives

INTERVENTIONS:
Other: Standard care encouraging family-mediated disclosure of hereditary cancer risk — At counseling, eligible at-risk relatives (who may benefit from disclosure of risk information) are listed on a specified protocol in collaboration between health care provider and the participant.
Other: Offer of health-care assisted disclosure by sending direct letters to at-risk relatives — The participant is offered that the health care provider at the cancer genetic unit mail a direct letter with personalized family risk information to all at-risk relatives that participant approve contact with.
  Arms: Intervention / Health-care assisted disclosure

SUMMARY:
This study evaluates if uptake of genetic counselling in high-risk families is increased when patients at cancer genetics clinics are being offered healthcare-assisted disclosure to at-risk relatives compared to current standard care (with family-mediated disclosure).

Patients/families who have undergone a cancer genetic investigation will be invited to participate in the study. All participants will receive standard care. Half of them will in addition be offered a healthcare-assisted disclosure with the service of direct letters to identified at-risk relatives distributed by the healthcare provider. After a year we will compare the proportion of at-risk relatives who have contacted a cancer genetic clinics in each study arm.

DETAILED DESCRIPTION:
(When the formal study protocol is published, this section will instead refer to the published study protocol).

This study is a multi-centre open label, prospective, randomized controlled superiority trial comparing an intervention of healthcare-assisted disclosure with standard care of family-mediated disclosure of hereditary cancer risk information in high-risk families in Sweden.

SUBJECTS AND METHODS

Patients/families will be enrolled and allocated in parallel to intervention or standard care.

All participants receive standard genetic counseling and information summarizing the results of their family investigation. They are informed about preventive measures when applicable, and are encouraged to inform their at-risk relatives (t=0 months).

The intervention component is the addition of a healthcare-assisted disclosure procedure. Participants in the intervention arm will be offered the service of sending letters directly to their at-risk relatives.

If the participant approves the offer, letters will be sent to eligible at-risk relatives deemed to be recommended genetic counseling within a year.

The direct letter will inform the at-risk relative that a cancer genetic investigation has been conducted in the family and the implications for him or her, and their blood relatives.

To facilitate access to further information, contact details to the closest cancer genetics unit are included in the letter. The letters are sent with registered mail in neutral envelopes which means that recipients will have to show proof of identity to retrieve the letter from their local delivery service provider.

METHODS FOR ASSESSMENT OF STUDY OUTCOMES

For participants in both study arms, contact details of the at-risk relatives are identified in collaboration between health care provider and the participant. The health care provider records the name, approximate or exact year of birth and postal address of each at-risk relative for follow-up.

At the time of follow-up (t=12 months) the research nurse will check whether the relatives, listed one year before, have contacted a Swedish cancer genetic unit. Primary outcome data is retrieved from the patient data registries at each clinic. The research nurse will also record additional data points from CRFs, enabling analysis of the other pre-specified outcome measures in the intervention arm.

The outcome data are reported back to the national study secretariat as plain numbers without any personal details of the at-risk relatives.

SAMPLE SIZE AND STATISTICAL METHODS

For sample size calculation and statistical methods, see attached documents.

INTERNAL PILOT, AUDIT and PROGRESS CRITERIA

As this protocol has never been tested in Swedish clinical practice an internal pilot phase is included in the outline of the project.

Progress criteria at each study site are evaluated at internal pilot point and thereafter at formal audit at least yearly. Internal pilot point is set to the time when 20 individuals in total (across the 3 pilot study sites) have been included and treated according to protocol.

Continuation of the full-powered study at the specific study site will be determined by considering the criteria filled, the potentially necessary amendments, and the degree of which the amendments deviate from the original piloted study protocol.

The outcomes and process criteria are found in the attached document.

ELIGIBILITY:
Inclusion criteria

1. Patient being offered a cancer genetic investigation for hereditary breast, ovarian or colorectal cancer.
2. Written consent to participate the study,
3. Belonging to a family with; a) familial breast cancer, b) familial colorectal cancer, c) pathogenic variant in PALB2, BRCA1/2 (Hereditary breast cancer, hereditary breast and ovarian cancer), MLH1, MSH2, MSH6, PMS2 (Lynch syndrome) and
4. Having at least one eligible at-risk relative (family member deemed to be an ARR recommended genetic counseling within a year).

Exclusion Criteria:

1. Cannot convey personal opinions and preferences by themselves.
2. No eligible at-risk relatives living in Sweden.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of genetic counselling among the patient's at-risk relatives | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Number of potential at-risk relatives who have contacted a Swedish cancer genetic unit out of the total number of potential at-risk relatives for each patient.

OTHER OUTCOMES:
Proportion of first-degree ARRs contacting a cancer genetics clinic | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Comparing intervention and control group with respect to proportion of first-degree ARRs who have contacted a Swedish cancer genetics clinic within 12 months of the proband receiving post-test genetic counselling because the proband is a carrier of a pathogenic variant in BRCA1, BRCA2, PALB2, MLH1, MSH2, MSH6, PMS2.
Proportion of distant ARRs contacting a cancer genetics clinic | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Comparing intervention and control group with respect to proportion of second-degree, third-degree or more distant ARRs who have contacted a Swedish cancer genetics clinic within 12 months of the proband receiving post-test genetic counselling because the proband is a carrier of a pathogenic variant in BRCA1, BRCA2, PALB2, MLH1, MSH2, MSH6, PMS2.
Intervention - Acceptance to offer (only intervention group) | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Number of potential at-risk relatives that proband allowed contact with, compared to total number of potential at-risk relatives for that specific patient. [proportion]
Intervention - Distribution of letters (only intervention group) | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Number of at-risk relatives that proband allowed contact with and where contact data allowed distribution of direct letter, compared to total number of potential at-risk relatives for that specific patient. [proportion]
Intervention - Collection of letters (only intervention group) | One year (12 months) following the first counselling session when implications of the cancer genetic investigation for the patient´s at-risk relatives is discussed, hence 12 months after t=0.
  Number of at-risk relatives that proband allowed contact with, contact data was sufficient and the registered letter was collected from the post-office within 12 months, compared to total number of potential at-risk relatives for that specific patient. [proportion]

CONTACTS AND LOCATIONS:
Locations (1):
- Cancergenetisk mottagning, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Access to aggregated data may be granted upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As requested by the publisher (peer reviewed journal).
Access Criteria: According to access to the peer reviewed journal.

REFERENCES:
- [Derived] Hawranek C, Ehrencrona H, Ofverholm A, Hellquist BN, Rosen A. Direct letters to relatives at risk of hereditary cancer-study protocol for a multi-center randomized controlled trial of healthcare-assisted versus family-mediated risk disclosure at Swedish cancer genetics clinics (DIRECT-study). Trials. 2023 Dec 17;24(1):810. doi: 10.1186/s13063-023-07829-5. PMID 38105176

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04197856/SAP_001.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04197856/ICF_002.pdf